CLINICAL TRIAL: NCT07337733
Title: Behavioral-Contextual Intervention for Emotional Regulation in Addictive Behaviors
Brief Title: Brief Contextual-Behavioral vs Twelve-Step Intervention for Emotion Regulation in Substance Use: Pilot Study
Acronym: MEX-BERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lauro Gutiérrez Castro (Other)
Responsible Party: Sponsor-Investigator, Lauro Gutiérrez Castro, Principal Investigator, Under The Tree Therapeutic Community
Organization: Under The Tree Therapeutic Community (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTT-PSI-MEX-BERA-001-2024
Record Dates: First submitted 2025-12-07; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders; Drug Use Disorder; Alcohol Use Disorder; Emotional Dysregulation; Distress Intolerance
Keywords: Emotion Regulation; Distress Tolerance; Substance Use Disorder; Behavioral Intervention; Psychological Flexibility
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study used a quasi-experimental, parallel-group design with matched allocation. Participants were assigned either to the Treatment Group, which received an 11-session behavioral-contextual intervention focused on emotion regulation and distress tolerance, or to the Comparison Group, which received usual residential care based on a 12-step model. Assessments were conducted at baseline and seven weeks later. The model emphasizes ecological validity within a therapeutic community setting, individual delivery of the intervention, and standardized procedures to ensure fidelity across sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral-Contextual Emotion Regulation Program (BCERP) (Experimental): Individual intervention comprising 11 weekly sessions (45 minutes each). The intervention combines functional ABC analysis, attentional focus training, crisis management skills (STOP protocol), distress tolerance training (DBT-SUD), mindfulness practices with behavioral anchoring, ACT techniques to enhance psychological flexibility, and consolidation exercises with relapse prevention.
  Interventions: Behavioral: Behavioral-Contextual Emotion Regulation Program (BCERP)
- Standard Residential Treatment Based on the Twelve-Step Facilitation Model (No Intervention): Standard therapeutic community residential program based on the 12-step model, without the structured sessions of the experimental protocol. Pre- and post-assessments applied at the same time points as the Treatment Group (TG).

INTERVENTIONS:
Behavioral: Behavioral-Contextual Emotion Regulation Program (BCERP) — The Behavioral-Contextual Emotion Regulation Program (BCERP) is a structured emotional regulation skills training intervention based on Applied Behavior Analysis principles and adapted to a therapeutic community setting for individuals undergoing substance use rehabilitation. Unlike interventions focused solely on psychoeducation, BCERP integrates intensive skills practice, gradual exposure to high-distress situations, and real-time feedback provided by trained therapists. The program includes modules on distress tolerance, behavioral restructuring, functional identification of emotions, and the strengthening of alternative, non-substance-related behaviors. BCERP is distinguished by its emphasis on continuous supervision, the use of contextual therapeutic language, and systematic progress monitoring through weekly behavioral indicators.
  Other Names: Behavioral-Contextual Intervention for Emotional Regulation in Addictive Behaviors; BCERP for Substance Use Rehabilitation
  Arms: Behavioral-Contextual Emotion Regulation Program (BCERP)

SUMMARY:
This study evaluated the effectiveness of a brief behavioral-contextual intervention delivered through 11 weekly individual sessions (45 minutes each) to improve emotion regulation, distress tolerance, and psychological flexibility among adults undergoing residential rehabilitation for problematic substance use in a Mexican therapeutic community. The intervention combined functional analysis, Dialectical Behavior Therapy strategies adapted for substance use disorders, and Acceptance and Commitment Therapy techniques. Participants received structured materials, including a session manual, mindfulness audio recordings, worksheets, and adapted behavioral monitoring tools.

A quasi-experimental pretest-posttest design with matched allocation was used. The Treatment Group (n = 19) received the structured intervention, while the Comparison Group (n = 17) received usual residential care based on a 12-step model. Primary assessments were administered at baseline and seven weeks after baseline. Primary outcome measures included changes in total scores on the Difficulties in Emotion Regulation Scale (DERS) and the Distress Tolerance Scale (DTS). Secondary outcomes included psychological flexibility (AAQ-II), emotion regulation strategies (ERQ reappraisal and suppression subscales), and behavioral indicators such as craving logs and engagement in value-consistent activities.

Procedures to ensure implementation fidelity included a standardized intervention manual, periodic clinical supervision, and consistent documentation using structured forms. Due to practical constraints and a moderate sample size, the statistical plan relied on robust analytical strategies, including nonparametric tests, permutation-based ANCOVA, and bootstrap estimation to evaluate effect sizes and sensitivity. All participants provided written informed consent, and the protocol was approved by an institutional ethics committee. Individual-level data will not be publicly shared due to confidentiality requirements; methodological materials and analytic scripts may be made available upon request and under confidentiality agreement.

DETAILED DESCRIPTION:
This study evaluated the effectiveness of a behavioral-contextual intervention, delivered in 11 weekly individual sessions (45 min each), aimed at improving emotion regulation, distress tolerance, and psychological flexibility among adults in residential rehabilitation for problematic substance use in a Mexican therapeutic community. The protocol combined functional analysis, DBT (SUD adaptations) and ACT techniques, practice materials (mindfulness audios, worksheets) and an adapted behavioral monitoring system. The design was quasi-experimental pre-post with a Treatment Group (TG; n = 19) and a Comparison Group (CG; n = 17) receiving usual care (12-step program). Primary measures were DERS, DTS, ERQ and AAQ-II administered at baseline and 7 weeks post-baseline. Implementation fidelity was supported by a manual, monthly supervision and standardized records. Analyses used robust methods (nonparametric tests, permutational ANCOVA, bootstrap, robust estimators).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Resident of the participating therapeutic community undergoing treatment for problematic substance use or alcohol.
* Capacity to provide informed consent and complete self-report assessments.

Exclusion Criteria:

* Active psychosis or unstable psychiatric comorbidity that precludes participation.
* Severe cognitive impairment preventing participation.
* Refusal to participate or unavailability to complete baseline and post assessments.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS-24 Total + Subscales) | Baseline to 7 weeks post-baseline
  The Difficulties in Emotion Regulation Scale - 24 item version (DERS-24), validated in Mexican populations, is a self-report measure assessing emotion regulation difficulties. The total score and five subscales are analyzed: Emotional Rejection, Emotional Dyscontrol, Emotional Interference, Emotional Inattention, and Emotional Confusion. Higher scores indicate greater difficulties in emotion regulation (worse outcome). Changes in total and subscale scores from baseline to post-intervention will be analyzed as continuous outcomes. No validated clinical cut-off scores exist; exploratory cohort analyses, when conducted, will use pre-specified sample-based thresholds (e.g., median or tertiles).
Distress Tolerance Scale (DTS) - Spanish Version | Baseline to 7 weeks post-baseline.
  Change in Distress Tolerance Scale (DTS) subscale scores - Tolerance, Appraisal, Absorption, Regulation. Change (Post - Pre) in DTS subscale scores. Subscale scoring (sum of items): Tolerance (3-15; higher = greater tolerance), Appraisal (6-30; higher = greater tolerance), Absorption (3-15; higher = greater tolerance), Regulation (3-15; higher = greater tolerance). Item 6 is reverse-scored.

SECONDARY OUTCOMES:
Emotion Regulation Questionnaire (ERQ) - Cognitive Reappraisal and Expressive Suppression Subscales | Baseline to 7 weeks.
  The Emotion Regulation Questionnaire (ERQ) is a 10-item self-report measure assessing habitual emotion regulation strategies. Two subscales are analyzed: Cognitive Reappraisal (6 items; score range 6-42), where higher scores indicate greater use of adaptive emotion regulation, and Expressive Suppression (4 items; score range 4-28), where higher scores indicate greater use of suppression, considered a less adaptive strategy. Primary analyses will examine continuous change in subscale scores from baseline to post-intervention. In secondary analyses, participants will be classified as responders or non-responders using a pre-specified cohort threshold defined as a change of at least 0.5 standard deviations from baseline (increase for reappraisal, decrease for suppression).
Acceptance and Action Questionnaire-II (AAQ-II) | Baseline to 7 weeks.
  The Acceptance and Action Questionnaire-II (AAQ-II) is a 7-item self-report measure assessing psychological flexibility and experiential avoidance. Total scores range from 7 to 49, with higher scores indicating greater experiential avoidance and lower psychological flexibility (worse outcome). Primary analyses will examine continuous change in total AAQ-II scores from baseline to post-intervention. In secondary analyses, participants will be classified as responders or non-responders using a pre-specified cohort threshold defined as a decrease of at least 0.5 standard deviations from baseline, indicating a clinically meaningful increase in psychological flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Lauro Gutiérrez Castro, Principal Investigator — Comunidad Terapéutica Under The Tree
Locations (1):
- Comunidad Terapéutica Under The Tree, Ajijic, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
If data sharing is conducted, only de-identified Individual Participant Data (IPD) will be made available, including coded demographic variables, baseline assessments, intervention adherence indicators, and pre-post outcome measures. No information that could directly or indirectly identify participants will be shared. Data will be provided exclusively for research purposes upon reasonable request and subject to a data-use agreement ensuring confidentiality and appropriate use. Study documentation such as manuals and analytic code may also be shared when relevant.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available only upon reasonable request from qualified researchers after completion of the primary analysis and publication of the study results. Availability will not include informed consent forms, as these documents are confidential and protected. The availability period will begin once the principal investigator receives a formal request and will remain open as long as there is a valid and ethically approved research purpose. All data will be provided in anonymized form and in full compliance with data protection regulations.
Access Criteria: Access to IPD and supporting information will be restricted to qualified researchers affiliated with academic or clinical institutions capable of meeting ethical and regulatory standards. Access will be limited to anonymized data relevant to clearly defined scientific research purposes approved by an ethics committee. Formal requests must be submitted to the principal investigator, who will evaluate the scientific rationale and confidentiality safeguards. Upon approval, data will be shared through a secure transfer mechanism under a data-use agreement that prohibits any attempt at re-identification.